CLINICAL TRIAL: NCT03817983
Title: Magnetic Resonance Enterography as a Screening Tool for Axial Spondyloarthritis in Crohn's Disease: A Prospective Single-center Cross-sectional Observational Study Using MRE Screening Followed by Clinical Assessment
Brief Title: MRE as a Screening Tool for axSpA in IBD
Acronym: ProSpA-CD
Status: Completed | Type: Observational
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Jobie Evans, Dr Jobie Evans (MD Student), Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: A094864
Record Dates: First submitted 2019-01-18; First posted 2019-01-28 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Axial Spondyloarthritis; Crohn Disease
MeSH Terms: conditions — Axial Spondyloarthritis; Crohn Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All subjects (cases and controls) will be asked to consent to provide research samples, including whole blood and stool, for storage and future analysis (serum for biomarker analysis, plasma for proteomic analysis, DNA for genotyping, and stool for microbiome analysis).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ProSpA-CD Screen Phase: MRE review for axSpA: Review of MRE scan for evidence of axSpA in Crohn's disease patients
  Interventions: Diagnostic Test: MRE review for evidence of axSpA in SIJs
- ProSpA-CD Assess Phase (cases): Clinical assessment and dedicated MRI of the spine and pelvis: Clinical assessment and dedicated MRI of the spine and pelvis to assess for evidence of axSpA for participants with abnormalities identified in the sacroiliac joints (SIJs) on MRE (cases).
  Interventions: Diagnostic Test: Clinical assessment and dedicated MRI of the spine and pelvis
- ProSpA-CD Assess Phase (controls): Clinical assessment and dedicated MRI of the spine and pelvis: Clinical assessment and dedicated MRI of the spine and pelvis to assess for evidence of axSpA for participants with normal SIJs (controls) on MRE.
  Interventions: Diagnostic Test: Clinical assessment and dedicated MRI of the spine and pelvis

INTERVENTIONS:
Diagnostic Test: MRE review for evidence of axSpA in SIJs — Screening for evidence of axSpA on the MRE scan of patients with Crohn's disease
  Groups: ProSpA-CD Screen Phase: MRE review for axSpA
Diagnostic Test: Clinical assessment and dedicated MRI of the spine and pelvis — Clinical assessment and dedicated MRI of the spine and pelvis to assess for evidence of axSpA
  Groups: ProSpA-CD Assess Phase (cases): Clinical assessment and dedicated MRI of the spine and pelvis; ProSpA-CD Assess Phase (controls): Clinical assessment and dedicated MRI of the spine and pelvis

SUMMARY:
This study aims to assess the effectiveness (specificity and sensitivity) of using magnetic resonance enterography (MRE) as a screening tool for axial spondyloarthritis (axSpA) in patients with Crohns disease. Patients with evidence of axSpA on MRE imaging will be assessed clinically for axSpA (including a dedicated axial magnetic resonance imaging scan of the spine and sacroiliac joints) and will be compared to a group of age and sex-matched control participants with Crohn's disease but with no evidence of axSpA on MRE imaging.

DETAILED DESCRIPTION:
Spondyloarthritis (SpA) is a term that encompasses psoriatic arthritis with axial disease, ankylosing spondylitis and non-radiological axial spondyloarthritis. The prevalence of SpA in the general population is estimated to be between 0.01%-2.5%. SpA patients have a high burden of inflammatory bowel disease (IBD), which primarily includes Crohn's disease (CD) and Ulcerative colitis (UC), with an estimated prevalence of 10%-12%. However, few studies have investigated the converse; the presence of IBD cases with undiagnosed SpA. Untreated SpA may lead to a significant impact on general health and quality of life; therefore early diagnosis and treatment is crucial. Most CD patients will have had a MRE assessment for their CD, which also captures the axial skeleton and can therefore be used to screen for evidence of axial SpA (axSpA). In this study, MRE images from consenting CD subjects will be reviewed for evidence of axSpA. CD patients with evidence of axSpA will then be reviewed in a rheumatology clinic to assess more specifically for SpA. This will include completion of patient reported outcome measures, clinical examination, routine blood tests, human leucocyte antigen (HLA)-B27 genotyping and a dedicated axial magnetic resonance imaging (MRI) scan. The patients will also be consented to participate in the second part of the study which will be to compare these 'cases' statistically to a 'control' group of age- and sex-matched CD subjects without MRE evidence of axSpA.

This study aims to: (i) determine the validity, sensitivity and specificity of MRE as a screening tool for axSpA in CD patients using dedicated axial MRI scans with clinical assessment as the gold standard; (ii) devise an algorithm of clinical indices that can be used as a screening tool for axSpA in CD cases.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are willing and able to give informed consent for participation in the study.
2. Male and female subjects aged 18 years or above.
3. Diagnosed by the gastroenterology team with Crohn's disease.
4. MRE imaging since 2015 for their Crohn's disease.

Exclusion Criteria:

1. Subjects unwilling or unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Crohn's disease (aged more than 18 years) who have had a MRE scan performed between January 1st 2015 and January 1st 2019
Sampling Method: Non-Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2020-08-08 (Actual); Study Completion 2020-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepak R Jadon, MBBCh PhD, Principal Investigator — CUH NHSFT
Locations (1):
- Rheumatology Research Unit, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- ProSpA-CD Screen Phase: MRE Review for Evidence of axSpA: Review of magnetic resonance enterography (MRE) imaging for evidence of axSpA in Crohn's disease patients
- ProSpA-CD Assess Phase (Cases): Clinical Assessment and Dedicated MRI of the Spine and Pelvis: Clinical assessment and dedicated MRI of the spine and pelvis to assess for evidence of axSpA for participants with abnormalities identified in SIJs (cases) on MRE.
- ProSpA-CD Assess Phase (Controls): Clinical Assessment and Dedicated MRI of the Spine and Pelvis: Clinical assessment and dedicated MRI of the spine and pelvis to assess for evidence of axSpA for participants with normal SIJs (cases) on MRE.
Period: ProSpA-CD Screen Phase
Arm/Group | ProSpA-CD Screen Phase: MRE Review for Evidence of axSpA | ProSpA-CD Assess Phase (Cases): Clinical Assessment and Dedicated MRI of the Spine and Pelvis | ProSpA-CD Assess Phase (Controls): Clinical Assessment and Dedicated MRI of the Spine and Pelvis
Started | 259 | 0 | 0
Completed | 259 (168/259 participants were recruited to the ProSpA-CD Assess phase of the study, of which 7/168 did not complete the study. In total, 161/259 participants completed the ProSpA-CD Assess phase.) | 0 | 0
Not Completed | 0 | 0 | 0
Period: ProSpA-CD Assess Phase
Arm/Group | ProSpA-CD Screen Phase: MRE Review for Evidence of axSpA | ProSpA-CD Assess Phase (Cases): Clinical Assessment and Dedicated MRI of the Spine and Pelvis | ProSpA-CD Assess Phase (Controls): Clinical Assessment and Dedicated MRI of the Spine and Pelvis
Started | 0 | 90 | 78
Completed | 0 | 90 | 71
Not Completed | 0 | 0 | 7
Not completed — MRI not performed | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- ProSpA-CD Assess Phase (Controls): Clinical Assessment and Dedicated MRI of the Spine and Pelvis: Clinical assessment and dedicated MRI of the spine and pelvis to assess for evidence of axSpA for participants with normal SIJs (controls) on MRE. Baseline data included for the 71 participants in this group that completed the study.
- ProSpA-CD Screen Phase: MRE Review for Evidence of axSpA Only: Review of MRE imaging of participants for evidence of axSpA changes. The 7 participants who started the ProSpA-CD Assess phase in the control group but did not complete the study are included in this group.
- Total: Total of all reporting groups
Arm/Group | ProSpA-CD Assess Phase (Cases): Clinical Assessment and Dedicated MRI of the Spine and Pelvis | ProSpA-CD Assess Phase (Controls): Clinical Assessment and Dedicated MRI of the Spine and Pelvis | ProSpA-CD Screen Phase: MRE Review for Evidence of axSpA Only | Total
Number analyzed (Participants) | 90 | 71 | 98 | 259
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 75 | 62 | 95 | 232
  >=65 years | 15 | 9 | 3 | 27
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 46.5 [35 to 56] | 43 [34 to 57] | 36 [29 to 45] | 41 [32 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 48 | 64 | 178
  Male | 24 | 23 | 34 | 81
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 90 | 71 | 98 | 259

OUTCOME MEASURES:

1. Primary Outcome: The Sensitivity and Specificity of MRE as a Screening Tool for Axial Spondyloarthritis in Crohn's Disease
Description: We assessed the SIJs on MRE imaging of patients with Crohn's disease (CD) for abnormalities potentially consistent with axial spondyloarthritis (axSpA), using a novel SIJ scoring system of 0-10 (0 = normal SIJs, 1-10 = abnormal SIJs). These patients were then assessed for evidence of axSpA using the Assessment of Spondyloarthritis International Society (ASAS) classification criteria for axSpA, including a dedicated axial MRI of the spine and pelvis. This primary outcome measure assessed the true positive rate (sensitivity) and true negative rate (specificity) of using MRE imaging of patients with CD to identify axSpA. A receiver operating characteristic (ROC) curve was generated using the novel SIJ scoring system of 0-10 and a 'diagnosis of axSpA' or 'no diagnosis of axSpA'. The ROC curve illustrated the true positive rate and true negative rate of using MRE as a screening tool for axSpA for each unit score (0-10) of the SIJ scoring system. This was performed using Stata 16 (2019).
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: Probability
Groups:
- ProSpA-CD Assess Phase (Cases + Controls): Clinical Assessment + Dedicated MRI of the Spine + Pelvis: Clinical assessment and dedicated MRI of the spine and pelvis to assess for evidence of axSpA for participants with abnormalities identified in SIJs (cases) and normal SIJs (controls) on MRE.
  The sensitivity, specificity and receiver operating characteristic curve of MRE as a screening tool for axSpA in Crohn's disease. Cases and control participants were combined for this statistical analysis.
Arm/Group | ProSpA-CD Assess Phase (Cases + Controls): Clinical Assessment + Dedicated MRI of the Spine + Pelvis
Number analyzed (Participants) | 161
Probability
  Sensitivity | 0.88 [0.69 to 0.98]
  Specificity | 0.50 [0.41 to 0.59]
  Area Under The Curve | 0.78 [0.65 to 0.86]

2. Secondary Outcome: The Number (and Percentage) of Participants With Evidence of Axial Spondyloarthritis on MRE Imaging Who Fulfill the 2009 ASAS Criteria for Axial Spondyloarthritis.
Description: Patients with Crohn's disease are at increased risk of developing axial spondyloarthritis (axSpA). MRE imaging is used to assess the extent of Crohn's disease in the small bowel and also captures the sacroiliac joints (SIJs), which are commonly affected in axSpA. The MRE images of participants with Crohn's disease were reviewed for abnormalities in the SIJs potentially consistent with axSpA. These participants were then clinically assessed for axSpA, ankylosing spondylitis (AS) and psoriatic arthritis (PsA). This included a clinical history and examination, blood tests (including HLA-B27 and inflammatory markers) and a dedicated axial MRI of the spine and pelvis. Radiographs of the SIJs, hands and feet were reviewed if available. The 2009 ASAS (Assessment of Spondyloarthritis International Society) classification criteria for axSpA, modified New York criteria for AS and classification for PsA (CASPAR) criteria were then used to classify patients with axSpA, AS and PsA respectively.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- ProSpA-CD Assess Phase (Cases): Clinical Assessment and Dedicated MRI of the Spine and Pelvis: Clinical assessment and dedicated MRI of the spine and pelvis to assess for evidence of axSpA for participants with abnormalities identified in SIJs (cases) on MRE.
  The number (and percentage) of participants with evidence of axial Spondyloarthritis on MRE imaging who fulfill the 2009 ASAS criteria for axial Spondyloarthritis.
Arm/Group | ProSpA-CD Assess Phase (Cases): Clinical Assessment and Dedicated MRI of the Spine and Pelvis
Number analyzed (Participants) | 90
Participants | 22

3. Secondary Outcome: The Number (and Percentage) of Participants With Evidence of Axial Spondyloarthritis on MRE Imaging Who Fulfill the Modified New York Criteria for Ankylosing Spondylitis
Description: as for outcome 2
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- ProSpA-CD Assess Phase (Cases): Clinical Assessment and Dedicated MRI of the Spine and Pelvis: Clinical assessment and dedicated MRI of the spine and pelvis to assess for evidence of axSpA for participants with abnormalities identified in SIJs (cases) on MRE.
  The number (and percentage) of participants with evidence of axial Spondyloarthritis on MRE imaging who fulfill the modified New York criteria for Ankylosing spondylitis
Arm/Group | ProSpA-CD Assess Phase (Cases): Clinical Assessment and Dedicated MRI of the Spine and Pelvis
Number analyzed (Participants) | 90
Participants | 8

4. Secondary Outcome: The Number (and Percentage) of Participants With Evidence of Axial Spondyloarthritis on MRE Imaging Who Fulfill the CASPAR Criteria for Psoriatic Arthritis
Description: as for outcome 2
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- ProSpA-CD Assess Phase (Cases): Clinical Assessment and Dedicated MRI of the Spine and Pelvis: Clinical assessment and dedicated MRI of the spine and pelvis to assess for evidence of axSpA for participants with abnormalities identified in SIJs (cases) on MRE.
  The number (and percentage) of participants with evidence of axial Spondyloarthritis on MRE imaging who fulfill the CASPAR criteria for psoriatic arthritis.
Arm/Group | ProSpA-CD Assess Phase (Cases): Clinical Assessment and Dedicated MRI of the Spine and Pelvis
Number analyzed (Participants) | 90
Participants | 8

5. Secondary Outcome: The Number (and Percentage) of Participants Fulfilling the 2009 ASAS Criteria for axSpA Proceeding to Non-pharmacological and Pharmacological Treatment of Their axSpA, as a Surrogate Measure of Change in Clinical Care as a Result of MRE Screening.
Description: This outcome measure focuses on the group of participants who fulfilled the 2009 ASAS classification criteria for axial spondyloarthritis in the ProSpA-CD Assess cases group. A total of 22 participants in the cases group fulfilled the 2009 ASAS classification criteria for axial spondyloarthritis (n=22/90).
Time Frame: 12 months
Population: This outcome measure focuses on the group of participants who fulfilled the 2009 ASAS classification criteria for axial spondyloarthritis in the ProSpA-CD Assess cases group. A total of 22 participants in the cases group fulfilled the 2009 ASAS classification criteria for axial spondyloarthritis (n=22/90).
Measure: Count of Participants; unit: Participants
Groups:
- ProSpA-CD Assess Phase (Cases): Clinical Assessment and Dedicated MRI of the Spine and Pelvis: Clinical assessment and dedicated MRI of the spine and pelvis to assess for evidence of axSpA for participants with abnormalities identified in SIJs (cases) on MRE.
  The number (and percentage) of participants fulfilling the 2009 ASAS classification criteria for axSpA proceeding to non-pharmacological and pharmacological treatment of their axSpA, as a surrogate measure of change in clinical care as a result of MRE screening.
Arm/Group | ProSpA-CD Assess Phase (Cases): Clinical Assessment and Dedicated MRI of the Spine and Pelvis
Number analyzed (Participants) | 22
Participants
  New Biologic Therapy | 4
  Non-Pharmacological Therapy | 5
  Continue Established Biological Therapy | 12
  Declined Treatment | 1

6. Secondary Outcome: The Predictive Value of Specific Extra-articular Features With a Diagnosis of Axial Spondyloarthritis in Crohn's Disease
Description: The MRE images of participants with Crohn's disease (CD) were reviewed for abnormalities in the SIJs potentially consistent with axSpA. The participants were then clinically assessed for axSpA, ankylosing spondylitis (AS) and psoriatic arthritis (PsA). The clinical assessment included age, sex, smoking status, alcohol consumption, occupation, site of CD, CD disease duration, history of extra-articular manifestations/ features, patient reported outcome measures, blood tests (including HLA B27 and inflammatory markers) and a dedicated axial MRI of the spine and pelvis. The 2009 ASAS (Assessment of Spondyloarthritis International Society) classification criteria for axSpA, modified New York criteria for AS and classification for PsA criteria were then used to classify patients with axSpA, AS and PsA respectively. Logistic regression analyses were performed to assess the association of extra-articular features and site of CD with a diagnosis of axSpA in CD, using Stata 16 (2019).
Time Frame: 12 months
Population: Logistic regression analysis for the association of extra-articular features (psoriasis, uveitis, erythema nodosum and orofacial granulomatosis) with axSpA in CD. Statistical significance level was set at 0.05.
Measure: Number (95% Confidence Interval); unit: Odds Ratio
Groups:
- ProSpA-CD Assess Phase (Cases): Clinical Assessment + Dedicated MRI of the Spine + Pelvis: Clinical assessment and dedicated MRI of the spine and pelvis to assess for evidence of axSpA for participants with abnormalities identified in SIJs (cases) on MRE.
  Logistic regression analysis of the association of extra-articular features (psoriasis, uveitis, erythema nodosum, pyoderma gangrenosum, orofacial granulomatosis and primary sclerosing cholangitis) with axSpA in Crohn's disease. Statistical significance level was set at 0.05.
Arm/Group | ProSpA-CD Assess Phase (Cases): Clinical Assessment + Dedicated MRI of the Spine + Pelvis
Number analyzed (Participants) | 90
Odds Ratio
  Psoriasis and axSpA: number analyzed (Participants) | 9
  Psoriasis and axSpA | 4.71 [1.14 to 19.46]
  Uveitis and axSpA: number analyzed (Participants) | 10
  Uveitis and axSpA | 3.71 [0.96 to 14.30]
  Erythema nodosum and axSpA: number analyzed (Participants) | 14
  Erythema nodosum and axSpA | 1.29 [0.36 to 4.61]
  Orofacial granulomatosis and axSpA: number analyzed (Participants) | 3
  Orofacial granulomatosis and axSpA | 1.57 [0.14 to 18.21]

7. Secondary Outcome: The Predictive Value of a Particular Site of Crohn's Disease (Colon, Ileum Etc) With a Diagnosis of Axial Spondyloarthritis in Crohn's Disease
Description: The MRE images of participants with Crohn's disease (CD) were reviewed for abnormalities in the SIJs potentially consistent with axSpA. The participants were then clinically assessed for axSpA, ankylosing spondylitis (AS) and psoriatic arthritis (PsA). The clinical assessment included age, sex, smoking status, site of CD, CD disease duration, history of extra-articular manifestations/ features, blood tests (including HLA B27 and inflammatory markers) and a dedicated axial MRI of the spine and pelvis. The 2009 ASAS (Assessment of Spondyloarthritis International Society) classification criteria for axSpA, modified New York criteria for AS and classification for PsA criteria were then used to classify patients with axSpA, AS and PsA respectively. Logistic regression analyses were performed to assess the association of extra-articular features and site of CD with a diagnosis of axSpA in CD, using Stata 16 (2019).
Time Frame: 12 months
Population: Logistic regression analysis for the association of the site of Crohn's disease (colon, ileum etc) with axSpA. Statistical significance level was set at 0.05.
Measure: Number (95% Confidence Interval); unit: Odds Ratio
Groups:
- ProSpA-CD Assess Phase (Cases): Clinical Assessment + Dedicated MRI of the Spine + Pelvis: Clinical assessment and dedicated MRI of the spine and pelvis to assess for evidence of axSpA for participants with abnormalities identified in SIJs (cases) on MRE.
  Logistic regression analysis for the association of the site of Crohn's disease with axSpA. Statistical significance level was set at 0.05.
Arm/Group | ProSpA-CD Assess Phase (Cases): Clinical Assessment + Dedicated MRI of the Spine + Pelvis
Number analyzed (Participants) | 90
Odds Ratio
  Ileal CD and axSpA: number analyzed (Participants) | 49
  Ileal CD and axSpA | 1.01 [0.38 to 2.64]
  Colonic CD and axSpA: number analyzed (Participants) | 10
  Colonic CD and axSpA | 1.38 [0.32 to 5.85]
  Ileocolonic CD and axSpA: number analyzed (Participants) | 31
  Ileocolonic CD and axSpA | 0.86 [0.31 to 2.39]

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- ProSpA-CD Screen Phase: MRE Review for Evidence of axSpA: Review of MRE imaging for evidence of axSpA in Crohn's disease patients.
Arm/Group | ProSpA-CD Screen Phase: MRE Review for Evidence of axSpA | ProSpA-CD Assess Phase (Cases): Clinical Assessment and Dedicated MRI of the Spine and Pelvis | ProSpA-CD Assess Phase (Controls): Clinical Assessment and Dedicated MRI of the Spine and Pelvis
All-Cause Mortality (participants affected / at risk) | 0/259 | 0/90 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/259 | 0/90 | 0/78
Other Adverse Events (participants affected / at risk) | 0/259 | 0/90 | 0/78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/83/NCT03817983/Prot_SAP_000.pdf